## Buprenorphine Plus Baclofen to Increase Analgesia in Healthy Volunteers

NCT04251819

November 14, 2025

## Statistical Analysis Plan

All baseline characteristics and outcome measures were analyzed descriptively. Specifically, the means and standard deviations within each group (i.e., Placebo, Baclofen 5mg, and Baclofen 10mg) were calculated for all continuous variables. For the baseline characteristic of age, the mean and standard deviation of the overall sample was also calculated. For the categorical variables, frequencies of each category within each group and in the overall sample were calculated. No analyses were conducted to compare the groups on any variable.